**Identifiers:** NCT03254550

**Unique Protocol ID:** Swazi PrEP study

**Brief Title:** PrEP Demonstration Study in Swaziland

**Date of document:** December 19<sup>th</sup> 2018

## Statistical analysis plan:

The data from the stepped-wedge randomized trial will be analyzed by first computing the number of clients who are initiated on PrEP at each healthcare facility in each of the 18 study months. We will then fit a negative binomial model that regresses the monthly number of clients who initiated PrEP onto a dichotomous indicator for the PPP phase (i.e., whether the healthcare facility was implementing the PPP in that month), study month as a continuous variable (whereby we will use fractional polynomials – with a maximum degree of two – to allow for non-linearities), and a facility-level fixed effect (i.e., a dichotomous indicator for each healthcare facility). The p-values for the point estimate for the intervention (i.e., the dichotomous indicator for the PPP phase) will be obtained using a non-parametric permutation test, which we will implement using the swpermute package in Stata.